CLINICAL TRIAL: NCT04421196
Title: Opioid-free Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Opioid-free Total Hip Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Currently does not have active IRB status.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00254474
Record Dates: First submitted 2020-05-19; First posted 2020-06-09 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-04

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard multimodal analgesic pathway with opioids (No Intervention): This is the control group, who will receive the current standard multimodal analgesic regimen, which includes opioids following total hip arthroplasty at Johns Hopkins Bayview Hospital.
  The current standard multimodal analgesic regimen utilizes the following medications: Gabapentin 300 mg, Celecoxib 200 mg (Meloxicam if sulfa), Opioid (fentanyl) & Non-opioid anesthetics (fluranes, propofol, ketamine, etc.); Periarticular injection: 0.25 % bupivacaine with epinephrine and Ketorolac IV; high volume cryotherapy, Ketorolac 30 mg IV, Oxycodone 5-10 mg PO, IV opioids (Morphine, hydromorphone), Acetaminophen 1000 mg PO q6hr
- Modified multimodal analgesic pathway without opioids (Experimental): This is the experimental group, who will receive a modified multimodal analgesic regimen, which excludes the use of any opioids.
  The modified multimodal analgesic regimen utilizes the following medications:
  includes the following medications: Gabapentin 300 mg, Celecoxib 200 mg (Meloxicam if sulfa), Non-opioid anesthetics (fluranes, propofol, ketamine, etc.); Periarticular injection: Liposomal bupivacaine, 0.25 % bupivacaine with epinephrine, Betamethasone sodium phosphate, betamethasone acetate and Ketorolac IV; high volume cryotherapy, Ketorolac 30 mg IV, Ketamine IV, Ketorolac 15 mg PO, Acetaminophen 1000 mg PO q6hr
  Interventions: Other: Exclusion of opioid analgesics

INTERVENTIONS:
Other: Exclusion of opioid analgesics — The intervention involves removing the option of patients having an opioid analgesic at any time point during the perioperative period.
  Arms: Modified multimodal analgesic pathway without opioids

SUMMARY:
The primary objective of investigators' proposed study is to demonstrate that the following two cohorts undergoing total hip arthroplasty will have equivalent visual analog scale (VAS) scores up to 3 months post-operatively: one that is administered a modified multimodal analgesic pathway without opioids and the other administered the current standard multimodal analgesic pathway used at Johns Hopkins Bayview Hospital (which includes opioids). The secondary objective is to demonstrate that these cohorts will also have equivalent functional outcomes as determined by both objective measures (such as hip range of motion) and patient-reported outcome measures, such as the Hip Disability and Osteoarthritis Outcome Score (HOOS) and the University of California at Los Angeles (UCLA) activity score.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages with end-stage primary hip osteoarthritis.

Exclusion Criteria:

* Patients with creatinine clearance between 30 and 60 mL/min
* Use of any opioid analgesics in the 6 months preceding surgery
* Revision total hip arthroplasty
* Patients with liver insufficiency
* Patients on chronic anticoagulation
* Workers compensation patients
* Patients who cannot receive Acetaminophen, Ketorolac, Celecoxib, or Gabapentin for any reason (e.g. allergies)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in post-operative pain assessed by the Visual analog scale (VAS) pain scores | From immediate post-operative period to 3 months post-operatively
  Post-operative pain scores ranging from 0 to 10; 0 being no pain and 10 being the worst pain ever felt

SECONDARY OUTCOMES:
Change in pain satisfaction as assessed by Hip Disability and Osteoarthritis Outcome Score (HOOS) | From pre-operative clinic visit to immediate post-operative period, then to 3 months post-operatively
  A patient-reported measure that assesses components such as assesses patient pain, satisfaction including stiffness and range of motion, activity limitations-daily living, sports and recreation function, and quality of life. Scores range from 0 to 100 with a score of 0 indicating the worst possible hip symptoms and 100 indicating no hip symptoms.
Change in Physical Activity level as assessed by the University of California at Los Angeles (UCLA) Scale | From pre-operative clinic visit to immediate post-operative period, and then to 3 months post-operatively
  The UCLA scale is a patient-reported measure ranging from 1 to 10. Patients indicate their most appropriate activity level, with 1 defined as "no physical activity, dependent on others" and 10 defined as "regular participation in impact sports."

CONTACTS AND LOCATIONS:
Overall Officials: Julius Oni, M.D., Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madras BK. The President's Commission on Combating Drug Addiction and the Opioid Crisis: Origins and Recommendations. Clin Pharmacol Ther. 2018 Jun;103(6):943-945. doi: 10.1002/cpt.1050. Epub 2018 Mar 23. PMID 29570781
- [Background] Rodriguez-Merchan EC, Vaquero-Picado A, Ruiz-Perez JS. Correction to: Opioid-Free Total Knee Arthroplasty? Local Infiltration Analgesia Plus Multimodal Blood-Loss Prevention Make it Possible. HSS J. 2019 Jul;15(2):209. doi: 10.1007/s11420-019-09679-x. Epub 2019 Apr 1. PMID 31327956
- [Background] Leas DP, Connor PM, Schiffern SC, D'Alessandro DF, Roberts KM, Hamid N. Opioid-free shoulder arthroplasty: a prospective study of a novel clinical care pathway. J Shoulder Elbow Surg. 2019 Sep;28(9):1716-1722. doi: 10.1016/j.jse.2019.01.013. Epub 2019 May 6. PMID 31072655
- [Background] Desmet M, Vermeylen K, Van Herreweghe I, Carlier L, Soetens F, Lambrecht S, Croes K, Pottel H, Van de Velde M. A Longitudinal Supra-Inguinal Fascia Iliaca Compartment Block Reduces Morphine Consumption After Total Hip Arthroplasty. Reg Anesth Pain Med. 2017 May/Jun;42(3):327-333. doi: 10.1097/AAP.0000000000000543. PMID 28059869
- [Background] Stevens RD, Van Gessel E, Flory N, Fournier R, Gamulin Z. Lumbar plexus block reduces pain and blood loss associated with total hip arthroplasty. Anesthesiology. 2000 Jul;93(1):115-21. doi: 10.1097/00000542-200007000-00021. PMID 10861154
- [Background] Becchi C, Al Malyan M, Coppini R, Campolo M, Magherini M, Boncinelli S. Opioid-free analgesia by continuous psoas compartment block after total hip arthroplasty. A randomized study. Eur J Anaesthesiol. 2008 May;25(5):418-23. doi: 10.1017/S026502150700302X. Epub 2007 Nov 21. PMID 18028577